CLINICAL TRIAL: NCT03965377
Title: Injuries Aren't Part of the Game: Developing an Injury Prevention Simulation Game to Better Engage Parents in Services
Brief Title: Developing an Injury Prevention Simulation Game to Better Engage Parents in Services -Home Safety Hero
Acronym: HSH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Sandra Azar, Professor, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00008278
Record Dates: First submitted 2019-04-10; First posted 2019-05-29 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Parenting
Keywords: effectiveness of gaming technology; knowledge of childhood injury prevention

STUDY DESIGN:
Intervention Model Description: teen parents and parents to be will be randomly assigned to game play (4 vs 1) to assess the effectiveness of the computer game to decrease time to identifying home hazards, improve identification of resolutions of hazards, and time to identify home hazards under distraction conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home Safety Hero game play (Experimental): Home Safety Hero is parental psychoeducational computer game to prevent childhood injuries
  Interventions: Behavioral: Home Safety Hero Computer Game

INTERVENTIONS:
Behavioral: Home Safety Hero Computer Game — Home Safety Hero computer game presents players with virtual rooms in a home where vilians have planted safety risks. It involves the player taking the role of a body guard for a child. It has three phases: 1. Identifying risks in a set of rooms (e.g., burn, falling, suffocation, poisoning); 2. Identifying risks and then selecting a resolution to reduce the risk or eliminate it entirely; and 3. Identifying risk when faced with distractions typical to home environments (e.g., phone ringing, fire engine siren sounds, a moving child).

SUMMARY:
This study will test the effectiveness of novel technology-based game to teach parents and parents to be home safety skills. These include the identification of home child injury risks under two conditions (with and without distraction) and how to resolve these risks to better protect preschool children from injuries. Few empirically validated home safety interventions exist and the best ones involve individual home visitors. These and others that use didactic instruction or provision of written material have poor response from low socioeconomic parents who are less literate and more resistant to outsiders entering their homes. The use of a computer game to provide education in this area is being tested for effectiveness and the game's engagement will also be examined.

Given cognitive problems in parents have been linked in the PI's work to child neglect (e.g., poor child supervision), links of performance on the game to cognitive capacities will also be examined in a preliminary way.

DETAILED DESCRIPTION:
The study will compare a group of parents and parents to be who play the game multiple times (n=15) to a wait list group (n=15) who just play it once. The study will examine reaction times to identification and resolution of the risks overall and by category of risk (e.g., poisoning, burns, suffocation, etc.). The study will also examine failures on levels of the game which are graded for difficulty. The game was designed for low failure rate to increase engagement and to improve motivation.

Changes in the participants' perception of efficacy in preventing injuries to children and their engagement with the game (using a standardized usability survey) will be examined. The study will also examine the role of experience with the use of technology and cognitive capacities in relation to performance and pre-post changes with multiple plays of the game.

ELIGIBILITY:
Inclusion Criteria:participants who are parents or parents to be from a high school program in Altoona, PA. For those less than age 18, parental permission for participation is required

-

Exclusion Criteria: non-English Speaking; ones whose due date falls in the study period and who are not likely to complete the project.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 30 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Learning | one week (four plays of the game) The outcomes average seconds until identification will be examined across the four game plays and also can be examined for each of four plays of the game.
  The game is designed to improve speed of identifying home safety hazards with and without distractions and also identify effective resolutions of the risks. Speed in identification is measured in seconds. Effectiveness in identifying resolutions is measured in seconds as well (e.g., seconds til correct response). Average time to identification of risks in each of the three phases of the game can be computed (Identification Phase, Resolution Phase, and Distraction Phase). The game will also give whether the resolutions selected are correct and thus, a percentage of correct resolutions can be computed for the entire resolution phase.

SECONDARY OUTCOMES:
:Perception of efficacy in preventing childhood injuries: PARENT SENSE OF INJURY COMPETENCE SCALE | pre and one week later This outcome will be measured using PARENT SENSE OF INJURY COMPETENCE SCALE. This instrument has 16 items that are rated on a 1-6 scale with 6 indicating greater efficacy. The items are totaled for overall efficacy perception.
  The participants' change in perception of efficacy in preventing childhood injuries
Engagement in the game | This instrument is collected one time at post test once they have completed game play. The time frame is one week after entering the study.
  A survey instrument [Usability Survey (UES)] will be collected that measures engagement in the game. This instrument has 26 items that assess engagement with the game rated on a five point scale from strongly disagree (1) to strongly agree (5). The ratings are totalled for an overall engagement score and this will be used to measure engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra T Azar, PhD, Principal Investigator — Penn State University
Locations (1):
- Sandra T. Azar, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No